CLINICAL TRIAL: NCT00284804
Title: An Open-label, Randomized, Multicenter, Phase II Study of MDX-060 in Combination With Gemcitabine, MDX060 in Combination With Dexamethasone, and Gemcitabine Monotherapy in Patients With Relapsed or Refractory Hodgkin's Disease
Brief Title: A Phase II Study of MDX-060 in Subjects With Relapsed or Refractory Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDX060-05/05E
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Hodgkin's Disease
Keywords: relapsed or refractory Hodgkin's Disease
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — iratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MDX-060 plus standard of care (Experimental): MDX-060 in combination with gemcitabine
  Interventions: Drug: MDX-060
- Standard of care (Active Comparator): Gemcitabine
  Interventions: Drug: MDX-060

INTERVENTIONS:
Drug: MDX-060 — anti-CD30 monoclonal antibody, i.v. weekly x 3 10 mg/kg
  Other Names: anti-CD30

SUMMARY:
This study is designed to determine the objective response rate in patients with relapsed or refractory Hodgkin's disease treated with MDX-060 in combination with gemcitabine or gemcitabine alone.

DETAILED DESCRIPTION:
Secondary objectives include:

* to characterize progression-free survival
* to characterize time to progression
* to determine response duration
* to characterize the effect of study drug on health-related quality of life
* to explore the correlation of positron emission tomography (PET) scan results with objective responses observed with conventional imaging in this patient population
* to characterize the immunogenicity response of MDX-060
* to characterize the safety of MDX-060, and
* to characterize the pharmacokinetic profile of MDX-060

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hodgkin's disease [HD] (excluding HIV-associated HD)
* Patients must have read, understood, and provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained
* Patients must have failed or relapsed following second line (i.e., salvage) chemotherapy or relapsed or failed following autologous stem cell transplant
* ECOG Performance Status of 0-2
* Patients must have bi-measurable disease
* At least 4 weeks since the last chemotherapy or radiation therapy with clinical evidence of recovery from any toxicity associated with such treatment
* Life expectancy 12 weeks or greater
* Screening laboratory values must be met
* Patients on corticosteroids must be tapered off the medication 2 weeks prior to study drug administration and remain off corticosteroids until study completion.

Exclusion Criteria:

* Previous treatment with any anti-CD30 antibody
* History of allogeneic transplant
* Any tumor lesion 10cm or greater in diameter
* Any other malignancy, excluding basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ. Any cancer from which the patient has been disease free for at least 5 years is permissible.
* Any significant active or chronic infection
* Apparent active or latent tuberculosis (TB) infection
* Patients who are pregnant or nursing
* Any underlying medical condition which, in the investigator's opinion, will make the administration of the study drug hazardous or obscure the interpretation of adverse events
* Concomitant chemotherapy, steroids, investigational agents, other anti-HD biologics, or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-11; Primary Completion 2008-05 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Day 50/57

SECONDARY OUTCOMES:
Progression-free survival | Day 50/57

CONTACTS AND LOCATIONS:
Overall Officials: Medarex Medical Monitor, Study Director — Medarex
Locations (17):
- United States (17):
  - City of Hope, National Medical Center, Duarte, California
  - California Oncology of the Central Valley, Fresno, California
  - University of California, San Diego/Moores UCSD Cancer Center, La Jolla, California
  - H. Lee Moffitt Cancer & Research Institute, Tampa, Florida
  - Rush Cancer Institute, Chicago, Illinois
  - St. Francis Hospital Center, Beech Grove, Indiana
  - American Health Network of Indiana, Indianapolis, Indiana
  - Division of Hematology/Oncology, Tufts-New England Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Nevada Cancer Institute, Las Vegas, Nevada
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - Mount Sinai School of Medicine, New York, New York
  - Carolina BioOncology Institute, PLLC, Huntersville, North Carolina
  - M.D. Anderson Cancer Center, The University of Texas, Houston, Texas
  - Mary Babb Randolph Cancer Center, Morgantown, West Virginia